CLINICAL TRIAL: NCT05218083
Title: REmotely Monitored, Mobile Health Supported Multidomain Rehabilitation Program With High Intensity Interval Training for COVID-19
Acronym: REMM-HIIT-CoV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Vanderbilt University Medical Center (Other); Ohio State University (Other); University of Kentucky (Other); University of Alabama at Birmingham (Other); Florida Atlantic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00109644; 1R01HD107103 (NIH)
Record Dates: First submitted 2022-01-06; First posted 2022-02-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Critical Illness; ICU Acquired Weakness; PICS; Cardiorespiratory Fitness
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REmotely Monitored, Mobile health supported Multidomain Rehabilitation Program with HIIT (Experimental): Patients will receive our REmotely monitored, Mobile health supported Multidomain Rehabilitation Program with High Intensity Interval Training Program (REMM-HIIT) with iWatch/iPhone.
  Interventions: Behavioral: REmotely monitored, Mobile health supported Multidomain Rehabilitation Program with High Intensity Interval Training (REMM-HIIT)
- Exercise education without personalized sessions or feedback (No Intervention): Patients will receive an exercise handout and iWatch/iPhone. Patients return home to exercise without personalized instruction and coaching.

INTERVENTIONS:
Behavioral: REmotely monitored, Mobile health supported Multidomain Rehabilitation Program with High Intensity Interval Training (REMM-HIIT) — REmotely Monitored, Mobile health-supported, High Intensity Interval Training consists of remotely monitored tailored, structured, progressive multidomain physical rehabilitation & personalized instruction & coaching.
  Patients complete 3 structured exercise sessions/week consisting of HIIT, strength, balance, and mobility exercises. Following warmup, patients increase workload at a heart rate corresponding to 95% VO2peak for 1-minute before returning to warm-up speed for 1-minute at a heart rate corresponding to 60% VO2peak.
  Strength includes functional strengthening exercises for lower extremities & general resistance exercises for major muscle groups.
  Balance incorporates static & dynamic exercises, including progressively narrowing base of support with eyes open or closed, reaching forward & backward starting within base of support & progressing to outside base of support.
  Mobility rehabilitation includes dynamic start/stop while walking and changing direction while walking.
  Arms: REmotely Monitored, Mobile health supported Multidomain Rehabilitation Program with HIIT

SUMMARY:
Multicenter, prospective, randomized controlled trial providing mobile health supported physical rehabilitation to 120 patients who have been critically ill with COVID-19 and who complete at least one exercise session.

DETAILED DESCRIPTION:
REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT) to improve recovery after hospital discharge in patients with COVID-19 will evaluate the feasibility of clinical-, physiological- and patient-centered outcomes associated with a remotely monitored, mobile health-supported high intensity interval rehabilitation exercise training to improve the functional recovery of survivors who have experienced critical illness with COVID-19 and have been discharged home from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of COVID-19 requiring hospital admission
* Discharged or expected to be discharged directly home from the hospital (not to a skilled nursing facility, inpatient rehabilitation center, or long-term acute care hospital)
* Able to ambulate with or without a gait aid prior to hospital discharge
* Age ≥ 18 years

Exclusion Criteria:

* Hospital discharge > 60 days unless readmitted to hospital in first 30 days, then 60 day window restarts and new exclusion is last hospital discharge > 60 days
* Not ambulating independently prior to COVID-19 illness (use of a gait aid permitted)
* Functional impairment resulting in inability to exercise at baseline
* Inability or unwillingness to comply with the study requirements or unable or unwilling to follow coaching via mobile-health iPhone interaction
* Any absolute contraindications to exercise, including but not limited to:

  * Recent (< 5 days) acute primary cardiac event
  * Unstable Angina
  * Uncontrolled dysrhythmias causing symptoms or hemodynamic compromise
  * Uncontrolled hypertension over 255 mmHg Systolic or 155 diastolic blood pressure
  * Symptomatic aortic stenosis
  * Uncontrolled symptomatic heart failure
  * Acute myocarditis or pericarditis
  * Suspected or known dissecting aneurysm
* Any adverse changes during GXT (i.e., persistent oxygen saturation drop below 88% while on prescribed oxygen therapy or significant hypotension such as mean arterial blood pressure < 60 mmHg on 2 consecutive readings within 1 minute)
* High risk for non-adherence as determined by screening evaluation
* Any condition, including cognitive impairment, that, in the judgment of the investigator, precludes participation because it could affect subject safety or ability of subject to complete the study
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minute walk distance | Baseline to 3 month follow-up
  distance walked in m

SECONDARY OUTCOMES:
Change in Cardiorespiratory fitness | Baseline to 3 month follow-up
  VO2P obtained during incremental Step Test
Change in physical function measured by Short Physical Performance Battery (SPPB) score. | Baseline to 3 month follow-up
  Scores range from 0 (frailty) to 12 (robustness).
Change in 30-sec sit to stand score | Baseline to 3 month follow-up
  Number of times the patient comes to a full standing position in 30 seconds
Change in Fried Frailty Index Score | Baseline to 3 month follow-up
  Score ranges from 0 (not frail) to 5 (frail).
Change in cognitive ability as measured by the MoCA Test | Baseline to 3 months follow-up
  Scores range from 0 to 30 with a lower score indicating more cognitive impairment.
Change in muscle mass obtained via MuscleSound | Baseline to 3 month follow-up
  Change in IMAT index as measured by MuscleSound
Compare EQ-5D-5L Score between intervention and control group | Baseline
  Scores range from -0.59 to where 1 is the best possible health state. Negative values represent health states perceived as worse than death, which is equal to 0
Compare EQ-5D-5L Score between intervention and control group | 3 month visit
  Scores range from -0.59 to where 1 is the best possible health state. Negative values represent health states perceived as worse than death, which is equal to 0
Compare EQ-5D-5L Score between intervention and control group | 6 month visit
  Scores range from -0.59 to where 1 is the best possible health state. Negative values represent health states perceived as worse than death, which is equal to 0
Compare Duke Activity Status Index (DASI) Score between intervention and control group | Baseline
  DASI scores range from 0 to 58.2, with a higher score indicating higher functional capacity.
Compare Duke Activity Status Index (DASI) Score between intervention and control group | 3 months
  DASI scores range from 0 to 58.2, with a higher score indicating higher functional capacity.
Compare Duke Activity Status Index (DASI) Score between intervention and control group | 6 months
  DASI scores range from 0 to 58.2, with a higher score indicating higher functional capacity.
Compare Lawton Score between intervention and control group | Baseline
  Score ranges from 0 (very dependent) to 8 (high function, independent)
Compare Lawton Score between intervention and control group | 3 months
  Score ranges from 0 (very dependent) to 8 (high function, independent)
Compare Lawton Score between intervention and control group | 6 months
  Score ranges from 0 (very dependent) to 8 (high function, independent)
Compare Hospital Anxiety and Depression Scale (HADS) Score between intervention and control group | Baseline
  Scores ranges from 0 to 21 for both anxiety and depression, with a higher score indicating more symptoms of depression or anxiety
Compare Hospital Anxiety and Depression Scale (HADS) Score between intervention and control group | 3 months
  Scores ranges from 0 to 21 for both anxiety and depression, with a higher score indicating more symptoms of depression or anxiety
Compare Hospital Anxiety and Depression Scale (HADS) Score between intervention and control group | 6 months
  Scores ranges from 0 to 21 for both anxiety and depression, with a higher score indicating more symptoms of depression or anxiety
Compare social determinants of health between intervention and control group | 3 months
  Completion of the Accountable Health Communities Health-Related Social Needs Screening Tool. A higher score indicates a higher Health-related social need.
Compare social determinants of health between intervention and control group | 6 months
  Completion of the Accountable Health Communities Health-Related Social Needs Screening Tool. A higher score indicates a higher Health-related social need.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, MD, Principal Investigator — Duke Clinical Research Institute
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Kentucky, Lexington, Kentucky
  - Duke University Health System, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No